CLINICAL TRIAL: NCT01703793
Title: A Parallel-group, Vehicle-controlled, Randomized, Double-blind Study of the Efficacy and Safety of Product 49778 and Product 10156 in Subjects With Seborrheic Dermatitis
Brief Title: Safety and Efficacy Study in Subjects With Seborrheic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicis Global Service Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP-1001-01
Record Dates: First submitted 2012-10-07; First posted 2012-10-11 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vehicle (Placebo Comparator): Vehicle (placebo) treatment, twice a week for four weeks.
  Interventions: Drug: Vehicle (placebo)
- Test Product 10156 (Experimental): Product 10156 treatment, twice a week for four weeks.
  Interventions: Drug: Test Product 10156
- Test Product 49778 (Experimental): Product 49778 treatment, twice a week for four weeks.
  Interventions: Drug: Test Product 49778

INTERVENTIONS:
Drug: Test Product 49778
  Arms: Test Product 49778
Drug: Test Product 10156
  Arms: Test Product 10156
Drug: Vehicle (placebo)
  Arms: Vehicle

SUMMARY:
The purpose of this study is to determine if two test products are safe and effective in the treatment of seborrheic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Investigator assessment of seborrheic dermatitis.
* Additional criteria as identified in the protocol.

Exclusion Criteria:

* History of or ongoing psoriasis of the scalp.
* History of or ongoing atopic dermatitis of the scalp.
* Additional criteria as identified in the protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Symptom Improvement (investigator assessment) | Week 4
  Proportion of subjects with a response of clear or almost clear, and at least a two-grade improvement from baseline to week 4

SECONDARY OUTCOMES:
Symptom Improvement (subject assessment) | Weeks 2 and 4
  Assess the change in the pruritus score from baseline to week 2 and to week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Lawrence, MD, Study Chair — Medicis Pharmaceutical
Locations (22):
- United States (22):
  - Fremont, California
  - Los Angeles, California
  - San Diego, California
  - New Haven, Connecticut
  - Aventura, Florida
  - Augusta, Georgia
  - Snellville, Georgia
  - Evansville, Indiana
  - Detroit, Michigan
  - Fridley, Minnesota
  - Paramus, New Jersey
  - Mount Kisco, New York
  - New York, New York
  - High Point, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Arlington, Texas
  - Austin, Texas
  - College Station, Texas
  - Plano, Texas
  - Webster, Texas
  - Salt Lake City, Utah